CLINICAL TRIAL: NCT06454786
Title: The Effect of Training Given by Simulation Method on the Self-confidence and Stress Levels of Nursing Students in Patient Intervention
Brief Title: The Effect of Simulation Method on Self-Confidence and Stress Levels in Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seher Yurt (Other)
Collaborators: Istanbul Kent University (Other)
Responsible Party: Sponsor-Investigator, Seher Yurt, Associated Professor, Istanbul Kent University
Organization: Istanbul Kent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IstanbulKentU-HEM-SY-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Simulation Training; Nursing Student; Self Confidence; Stress
Keywords: Simulation Training; Nursing Student; Self Confidence; Stress

STUDY DESIGN:
Intervention Model Description: Two groups with experimental and control groups
Who Masked: Outcomes Assessor
Masking Description: In order to prevent selection bias in the study, the assignment to the experimental and control groups will be made on a computer by a person who is unfamiliar with the research process. The analysis of the data will be done by a statistics expert who is outside the research process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simülation intervention group (Experimental): The Student Diagnosis Form, Self-Confidence/Efficacy Scale in Patient Intervention and Perceived Stress Scale will be applied first to this group. Then, face-to-face theoretical training will be given. Following the theoretical training, simulation training will be given in the Simulation Laboratory in line with the Nursing Care Scenario in Cardiogenic Shock. Simulation training will be conducted in 10 groups of 5 people and will be completed in 2 days. Each student in the group will actively participate in the simulation training within the scope of their role in the scenario. Posttests will be administered to both groups 2 weeks after the simulation training.
  Interventions: Other: Simulation Method
- Control group (No Intervention): The Student Diagnosis Form, Self-Confidence/Efficacy Scale in Patient Intervention and Perceived Stress Scale will be applied first to this group. Then, face-to-face theoretical training will be given. Post-tests will be administered 2 weeks after the theoretical training.

INTERVENTIONS:
Other: Simulation Method — Management of cardiogenic shock scenario on an advanced simulation mannequin
  Arms: simülation intervention group

SUMMARY:
The aim of this study was to determine the impact of training provided through simulation method on self-confidence and stress levels in nursing students during patient intervention.

DETAILED DESCRIPTION:
Improving nursing students' clinical skills and enhancing their professional competencies by increasing their patient intervention skills and strengthening their ability to cope with stress is crucial. High professional confidence among nursing students is fundamental to providing effective patient care, which is critical for patient safety and satisfaction. Simulation training is an effective tool used to enhance nursing students' practical experiences in clinical settings. This method provides students with the opportunity to encounter real-life scenarios in a controlled environment and intervene in these situations. Additionally, simulation training can help develop coping skills for dealing with stress, as it prepares students for situations they may encounter in real clinical settings. The aim of this study is to determine the impact of training provided through simulation method on self-confidence and stress levels in nursing students during patient intervention.

The students included in the study will be divided into experimental and control groups through full randomization. The Student Identification Form will be administered to both groups initially. The theoretical part of Shock Nursing Care (SNC) training will be provided to the control group through in-class face-to-face education. Following the theoretical training, skills training will be conducted in the nursing skills laboratory using the demonstration method. Students will be evaluated using the Self-Confidence/Competence in Patient Intervention Scale and the Perceived Stress Scale before and after the training. The study group will receive theoretical education similarly to the control group through in-class face-to-face education. Following the theoretical education, simulation training will be conducted in the Simulation Laboratory based on the SNC Scenario. Simulation training will be conducted in groups of 10, consisting of 5 students each. Each student will be provided the SNC scenario to practice. Students will be evaluated using the Self-Confidence/Competence in Patient Intervention Scale and the Perceived Stress Scale before and after the training. The mean scores of both groups on the Self-Confidence/Competence in Patient Intervention Scale and the Perceived Stress Scale will be compared both between and within groups. Pre-graduation nursing simulation education will contribute to enhancing students' patient intervention skills and stress coping abilities.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research, being a senior nursing student

Exclusion Criteria:

* Not participating in any simulation training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Self-Confidence/Efficacy Scale in Patient Intervention | Pre-test, post-test (2nd weeks later)
  The scale developed for health professional students with scenario-based simulation-based teaching experience includes 18 items and is evaluated according to a 5-point Likert system (1 = Strongly Disagree, 2 = Disagree, 3 = Undecided, 4 = Agree, 5 = Strongly Agree). While a high score means confidence, a low score means lack of self-confidence in students. Therefore, in clinical practice, the highest possible score is 55 and the lowest score is 11.

SECONDARY OUTCOMES:
Perceived Stress Scale for Nursing | Pre-test, post-test (2nd weeks later)
  The scale consists of 29 items and measures perceived stress for nursing.

CONTACTS AND LOCATIONS:
Overall Officials: SEHER YURT, Principal Investigator — Istanbul Kent University
Locations (1):
- Istanbul Kent University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No